CLINICAL TRIAL: NCT02644720
Title: Neural Compensation, Visual Function and Visual Quality in Senile Cataract Patients After Monofocal or Multifocal Intraocular Lens Implantation
Brief Title: Neural Compensation, Visual Function and Visual Quality After Monofocal or Multifocal Intraocular Lens Implantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Professor in Childhood Cataract Program of the Chinese Ministry of Health(CCPMOH), Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCPMOH2010-China12
Record Dates: First submitted 2015-12-27; First posted 2016-01-01 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Dexamethasone; Multifocal Intraocular Lenses

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- multifocal intraocular lens group (Experimental)
  Interventions: Procedure: multifocal intraocular lens implantation; Drug: Dexamethasone; Device: multifocal intraocular lens (IOL) (Tecnis ZMB00)
- monofocal intraocular lens group (Active Comparator)
  Interventions: Procedure: monofocal intraocular lens implantation; Drug: Dexamethasone; Device: monofocal intraocular lens (IOL) (Tecnis ZCB)

INTERVENTIONS:
Procedure: multifocal intraocular lens implantation — In this group, the surgery was performed with cataract extraction and multifocal intraocular lens (IOL) (Tecnis ZMB00). The standard technique in all patients consisted of sutureless phacomulsifacation using the Legacy 2000 Series and Infinity phacoemulsification machine (Alcon Laboratories Inc., Fort Worth, Texas, USA), with clear corneal incisions up to 3.2 mm and 5.0 to 5.5 mm capsulorhexis. Surgery in the fellow eye was performed 1 month later in each patient.
  Arms: multifocal intraocular lens group
Procedure: monofocal intraocular lens implantation — In the group, the surgery was performed with cataract extraction and monofocal intraocular lens (IOL) (Tecnis ZCB). The surgery technique was same as the multifocal intraocular lens group
  Arms: monofocal intraocular lens group
Drug: Dexamethasone — All patients received subconjunctival dexamethasone (2 mg) during surgery
Device: multifocal intraocular lens (IOL) (Tecnis ZMB00)
  Arms: multifocal intraocular lens group
Device: monofocal intraocular lens (IOL) (Tecnis ZCB)
  Arms: monofocal intraocular lens group

SUMMARY:
Multifocal intraocular lenses (MIOLs) provide enhanced far and near visual acuity, but they can bring about halos and glare, which are caused by design deficiencies of the IOLs. Compared to monofocal intraocular lens, pseudo accommodation in nonphysiological state may increase the difficulty of neural compensation reconstruction in patients with multifocal intraocular lens implantation. Patients enrolled into the study will be followed for 1 year and will have study visits preoperatively, at 1 week, 3 months, 6 months, 12 months postoperatively.In this trial, we aimed to specify the time of neural compensation reconstruction in patients and to explore the changes of visual function in senile patients with monofocal or multifocal intraocular lens implantation.

DETAILED DESCRIPTION:
Cataract extraction and intraocular lens (IOL) implantation are the current standard treatments for age-related cataract (ARC). Cataract surgery increases visual acuity but may lead to complaints after surgery. Multifocal intraocular lenses (MIOLs) provide enhanced far and near visual acuity, but they can bring about halos and glare, which are caused by design deficiencies of the IOLs. Fortunately, most of the halos and glare diminish with time. Niels et al noted that neural adaptation (NA) may explain the lower incidence of glare and halos in their study. Compared to monofocal intraocular lens, pseudo accommodation in nonphysiological state may increase the difficulty of neural compensation reconstruction in patients with multifocal intraocular lens implantation.

In the present study, the investigators evaluated the activity of neurons in the visual cortex using fMRI both preoperatively and postoperatively. In addition, the investigators evaluated postoperative changes in VF, including visual acuity (VA), contrast sensitivity (CS), straylight values (SVs), and pattern visual evoked potential (PVEP), stereoscopic vision, wavefront aberrations at 1 week, 3 months, 6 months, 12 months postoperatively.In this trial, the investigators aimed to specify the time of neural compensation reconstruction in patients and to explore the changes of visual function in senile patients with monofocal or multifocal intraocular lens implantation.

ELIGIBILITY:
Inclusion Criteria:

* visual acuity less than 0.3
* Cataracts in both eyes classified by the Lens Opacity Classification System III
* Corneal astigmatism less than 1.5 diopters (D)
* Capability of understanding and signing the informed consent

Exclusion Criteria:

* Corneal astigmatism ≥ 1.5D.
* History of neurological or psychiatric disorders; systemic disease such as severe hypertension or diabetes mellitus that might interfere with the visual outcomes.
* Associated ocular disease that could interfere with final results
* Previous anterior and posterior segment surgery and intraoperative or postoperative complications
* Driving at night frequently; excessive expectations for visual outcomes

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-01; Primary Completion 2019-01 (Estimated); Study Completion 2019-01

PRIMARY OUTCOMES:
Change from contrast sensitivity | 1 week, 1 month, 3 month, 6 month,1 year after surgery
  Contrast sensitivity (CS) was tested with a Contrast Glare Tester 1000
Change from functional magnetic resonance imaging | 1 week, 1 month, 3 month, 6 month,1 year after surgery

SECONDARY OUTCOMES:
Change from best corrected visual acuity | 1 week, 1 month, 3 month, 6 month,1 year after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Weirong Chen, M.D., Study Director — Zhongshan Ophthalmic Center, Sun Yat-sen University; Yizhi Liu, M.D.;Ph.D., Study Chair — Zhongshan Ophthalmic Center, Sun Yat-sen University; Haotian Lin, M.D.;Ph.D., Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhognshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Yao K, Bao Y, Ye J, Lu Y, Bi H, Tang X, Zhao Y, Zhang J, Yang J. Efficacy of 1% carboxymethylcellulose sodium for treating dry eye after phacoemulsification: results from a multicenter, open-label, randomized, controlled study. BMC Ophthalmol. 2015 Mar 20;15:28. doi: 10.1186/s12886-015-0005-3. PMID 25880685
- [Background] Kalantzis G, Papaconstantinou D, Karagiannis D, Koutsandrea C, Stavropoulou D, Georgalas I. Post-cataract surgery diplopia: aetiology, management and prevention. Clin Exp Optom. 2014 Sep;97(5):407-10. doi: 10.1111/cxo.12197. PMID 25138745
- [Background] Hayashi K, Hayashi H, Nakao F, Hayashi F. Correlation between pupillary size and intraocular lens decentration and visual acuity of a zonal-progressive multifocal lens and a monofocal lens. Ophthalmology. 2001 Nov;108(11):2011-7. doi: 10.1016/s0161-6420(01)00756-4. PMID 11713071
- [Background] Kim MJ, Zheleznyak L, Macrae S, Tchah H, Yoon G. Objective evaluation of through-focus optical performance of presbyopia-correcting intraocular lenses using an optical bench system. J Cataract Refract Surg. 2011 Jul;37(7):1305-12. doi: 10.1016/j.jcrs.2011.03.033. PMID 21700107
- [Background] Pieh S, Lackner B, Hanselmayer G, Zohrer R, Sticker M, Weghaupt H, Fercher A, Skorpik C. Halo size under distance and near conditions in refractive multifocal intraocular lenses. Br J Ophthalmol. 2001 Jul;85(7):816-21. doi: 10.1136/bjo.85.7.816. PMID 11423456
- [Derived] Lin H, Zhang L, Lin D, Chen W, Zhu Y, Chen C, Chan KC, Liu Y, Chen W. Visual Restoration after Cataract Surgery Promotes Functional and Structural Brain Recovery. EBioMedicine. 2018 Apr;30:52-61. doi: 10.1016/j.ebiom.2018.03.002. Epub 2018 Mar 7. PMID 29548900
- See also: Description Home page of Zhongshan Ophthalmic Center — http://www.gzzoc.com/